CLINICAL TRIAL: NCT03740464
Title: Long-acting Granulocyte Colony Stimulating Factor for the Prevention Febrile Neutropenia in Epithelial Ovarian Cancer: A Phase 3 Randomized Control Study
Brief Title: Long-acting G-CSF for Febrile Neutropenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EOC-GCSF
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Epithelial Ovarian Cancer; Colony Stimulating Factors; Febrile Neutropenia; Myelosuppression Adult; Adverse Event; Cost-effectiveness
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Febrile Neutropenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients in study group accept long-acting granulocyte colony stimulating factor 48 hours from the chemotherapy and regular interventions for myelosuppression.
  Interventions: Drug: long-acting granulocyte colony stimulating factor; Drug: Short-term granulocyte colony stimulating factor
- Control group (Active Comparator): Patients in control group only accept regular interventions for myelosuppression rather than long-acting granulocyte colony stimulating factor.
  Interventions: Drug: Short-term granulocyte colony stimulating factor

INTERVENTIONS:
Drug: long-acting granulocyte colony stimulating factor — A 6 mg of polyethylene glycol granulocyte colony stimulating factor will be given to patients of study group
  Other Names: polyethylene glycol granulocyte colony stimulating factor
  Arms: Study group
Drug: Short-term granulocyte colony stimulating factor — Short-term granulocyte colony stimulating factor will be given to all patients according to the severity of myelosuppression

SUMMARY:
This study aims to analyze the effects of long-acting granulocyte colony stimulating factor (G-CSF) on the prevention febrile neutropenia (FN) in epithelial ovarian cancer. Patients are randomized into study group and control group. In study group, patients accept long-acting G-CSF 48 hours from the chemotherapy. While the control group accept regular treatment rather than long-acting G-CSF. The primary end is the incidence of FN in every course of chemotherapy. The secondary ends include: the incidences of myelosuppression, doses of G-CSF and its expenses, visits to outpatient and emergency clinics, adverse events related to G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Willing to accepted debulking surgeries and adjuvant chemotherapy
* Good performance status
* Aged 18 years or older
* Signed an approved informed consents
* No immunosuppressive disease

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
febrile neutropenia | One year
  the incidence of febrile neutropenia happened during each course of chemotherapy

SECONDARY OUTCOMES:
myelosuppression | One year
  the incidence of the incidence of febrile neutropenia happened during each course of chemotherapy happened during each course of chemotherapy
doses of granulocyte colony stimulating factor | One year
  total doses of all granulocyte colony stimulating factor
expenses of granulocyte colony stimulating factor | One year
  total expenses of all granulocyte colony stimulating factor
visits to the hospital | One years
  visits to outpatient and emergency clinics
adverse events | One year
  adverse events related to G-CSF according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03
progression-free survival | Five years
  progression-free survival after the primary treatment of ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li L, Ma S, Wu M, Tan X, Zhong S, Lang J. The prophylactic effects of long-acting granulocyte colony-stimulating factor for febrile neutropenia in newly diagnosed patients with epithelial ovarian cancer: a randomised controlled study. BMJ Support Palliat Care. 2019 Dec;9(4):373-380. doi: 10.1136/bmjspcare-2019-001862. Epub 2019 Aug 29. PMID 31467066